CLINICAL TRIAL: NCT00086762
Title: Chemotherapy and Mindfulness Relaxation: A Randomized Trial at M.D. Anderson Cancer Center and M.D. Anderson Community Clinical Oncology Program
Brief Title: Mindfulness Relaxation Compared With Relaxing Music and Standard Symptom Management Education in Treating Patients Who Are Undergoing Chemotherapy For Newly Diagnosed Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2004-0024; MDA-CCC-0106; CDR0000357213 (Other: NCI); NCI-2009-00860 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific; Breast Cancer; Gastrointestinal Cancer; Disease (or Disorder); Gynecological; Prostate Cancer
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific; mindfulness relaxation
MeSH Terms: conditions — Vomiting; Breast Neoplasms; Gastrointestinal Neoplasms; Disease; Prostatic Neoplasms; Nausea | interventions — Therapeutics; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MR Therapy (Experimental): Participants receive Mindfulness Relaxation (MR) therapy as in the pilot phase. A CD with the mindfulness relaxation technique recorded on it will be given to participant. Participant to listen to the recording for about 30 minutes before receiving chemotherapy and during the time they are receiving chemotherapy. In addition to the mindfulness relaxation technique, they will also receive general information about how to manage symptoms that develop due to the chemotherapy they are receiving.
  Interventions: Behavioral: MR Therapy; Behavioral: Questionnaires
- Relaxing Music (RM) Therapy (Experimental): Arm II: Participants listen to relaxing music (with no instructions on relaxation techniques) for 30 minutes before and during each chemotherapy session AND at least once daily for the entire duration of chemotherapy treatment.
  Interventions: Behavioral: Relaxing Music (RM) Therapy; Behavioral: Questionnaires
- Standard Symptom Management (Active Comparator): Arm III: Participants receive standard symptom management education.
  Interventions: Behavioral: Standard Symptom Management; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: MR Therapy — Arm I: Participants receive Mindfulness Relaxation (MR) therapy as in the pilot phase. Instructions given on breathing techniques and other practices to help relax mind and body.
  Arms: MR Therapy
Behavioral: Relaxing Music (RM) Therapy — Participants listen to relaxing music (with no instructions on relaxation techniques) for 30 minutes before and during each chemotherapy session AND at least once daily for the entire duration of chemotherapy treatment
  Arms: Relaxing Music (RM) Therapy
Behavioral: Standard Symptom Management — Participants receive standard symptom management education. General information received about how to manage symptoms that develop due to the chemotherapy.
  Arms: Standard Symptom Management
Behavioral: Questionnaires — Questionnaire completion at baseline, during the middle of chemotherapy treatment, and at chemotherapy completion.
  Other Names: surveys

SUMMARY:
RATIONALE: Mindfulness relaxation, a technique to help patients quiet their thoughts and relax their bodies before and during chemotherapy, may reduce or prevent nausea and vomiting. It may also help improve mental health, quality of life, and immune function in patients receiving chemotherapy.

PURPOSE: This randomized clinical trial is studying mindfulness relaxation to see how well it works compared to relaxing music or standard symptom management education in treating patients who are receiving chemotherapy for newly diagnosed solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of mindfulness relaxation vs relaxing music vs standard symptom management education on conditioned and nonconditioned nausea and vomiting in patients with newly diagnosed solid tumors undergoing chemotherapy.

Secondary

* Compare mental health (anxiety, depression, and distress), quality of life (cancer-related symptoms, fatigue, sleep, and pain), and immune function in patients receiving these interventions.

OUTLINE: This is a multicenter study comprising a pilot phase followed by a randomized phase. (Pilot phase completed as of 3/10/2012.)

* Pilot phase: Patients undergo mindfulness relaxation (MR) therapy comprising listening to instructions on breathing techniques and other mind and body relaxation practices on compact disc for 30 minutes before and during each chemotherapy session AND at least once daily for the entire duration of chemotherapy treatment. (Pilot phase completed as of 3/10/2012.)
* Randomized phase: Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients undergo MR therapy as in the pilot phase.
  * Arm II: Patients listen to relaxing music (with no instructions on relaxation techniques) for 30 minutes before and during each chemotherapy session AND at least once daily for the entire duration of chemotherapy treatment.
  * Arm III: Patients receive standard symptom management education. In both phases, nausea and vomiting, mental health (anxiety, depression, and distress), and quality of life (cancer-related symptoms, fatigue, sleep, and pain) are assessed at baseline, periodically during treatment, and then at 3 months.

Patients are followed annually for up to 5 years for survival.

PROJECTED ACCRUAL: A total of 474 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. are >/= 18 years of age
2. are anticipated to undergo at least four cycles of chemotherapy treatment
3. have had no previous treatment with chemotherapy
4. have no evidence of distant metastatic disease
5. can read/speak in English or Spanish
6. have no known psychotic diagnosis
7. have an expected survival of at least 6 months

Exclusion Criteria:

1. have a known psychotic diagnosis
2. will undergo an undefined number of chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2004-06 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Conditioned nausea and vomiting as measured by Morrow assessment of nausea and emesis (MANE) | Up to 12 months post treatment
  Number of incidents conditioned nausea and vomiting as measured by MANE at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment
Distress as measured by Impact of Event Scale (IES) | Up to 12 months post treatment
  Distress as measured by Impact of Event Scale (IES) at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment
Fatigue as measured by brief fatigue inventory (BFI) | Up to 12 months post treatment
  Fatigue as measured by brief fatigue inventory (BFI) at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment
Anxiety as measured by Spielberger State/Trait Anxiety Scale (STAI) | Up to 12 months post treatment
  Anxiety as measured by Spielberger State/Trait Anxiety Scale (STAI) at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment
Depression as measured by Center for Epidemiology-Depression (CES-D) | Up to 12 months post treatment
  Depression as measured by Center for Epidemiology-Depression (CES-D) at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment.
Sleep as measured by Pittsburgh Sleep Quality Index (PSQI) | Up to 12 months post treatment
  Sleep as measured by Pittsburgh Sleep Quality Index (PSQI) at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment
Pain as measured by brief pain inventory (BPI) | Up to 12 months post treatment
  Pain as measured by brief pain inventory (BPI) at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment
Quality of life as measured by Functional Assessment of Cancer Therapy | Up to 12 months post treatment
  Quality of life as measured by Functional Assessment of Cancer Therapy at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment

SECONDARY OUTCOMES:
Immune suppression as measured by cytotoxicity, stimulated release of IL-12, -4, -10, intracellular cytokines and lymphocyte phenotype | Up to 12 months post treatment
  Immune suppression as measured by cytotoxicity, stimulated release of IL-12, -4, -10, intracellular cytokines and lymphocyte phenotype at baseline, after course 2 or 3, at end of treatment, and then 6 and 12 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jon Hunter, MD, FRCP, Principal Investigator — Mount Sinai Hospital, Canada; Lorenzo Cohen, PHD, Study Chair — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - University of Texas M.D. Anderson CCOP Research Base, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin